CLINICAL TRIAL: NCT06720337
Title: Comparative Study Between the Analgesic Effect of Dexmedetomidine and Magnesium Sulfate As Adjuvant to Bupivacaine Using Ultrasound-Guided Transversus Abdominis Plane Block in Abdominal Hysterectomy : a Randomized Double-blinded Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mahfouz Ali, resident doctor at Anaesthesia, Intensive Care and Pain Management department Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dexmedetomidine and Mgso4 TAP
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Hysterectomy
Keywords: ultrasound-Guided Transversus Abdominis Plane Block
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly allocated into one of the two study designed groups using computer-generated random numbers table.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group A (Experimental): Patients will receive 18 ml 0.5% bupivacaine (Sunnypivacaine®) plus 0.5 µg/kg of dexmedetomidine (Precedex® 100 µg/ml) diluted in 2 ml of normal saline at each side
  Interventions: Drug: bupivacaine 0.5%; Drug: Dexmedetomidine
- group b (Experimental): patients will receive 18 ml 0.5% bupivacaine (Sunnypivacaine®) plus 1.5 mL (150 mg) MgSO4 and 0.5 mL normal saline at each side
  Interventions: Drug: bupivacaine 0.5%; Drug: MgSO4

INTERVENTIONS:
Drug: bupivacaine 0.5% — patients will receive 18 ml 0.5% bupivacaine (Sunnypivacaine®) using Ultrasound-Guided TAP Block Technique
Drug: Dexmedetomidine — patients will receive plus 0.5 µg/kg of dexmedetomidine (Precedex® 100 µg/ml) diluted in 2 ml of normal saline at each side
  Arms: group A
Drug: MgSO4 — patients will receive plus 1.5 mL (150 mg) MgSO4 and 0.5 mL normal saline at each side
  Arms: group b

SUMMARY:
Over 80% of patients who undergo surgery suffer from acute postoperative pain, with 75% of them rating the pain severity as moderate, severe, or extreme. Studies have shown that less than 50% of patients who undergo surgery report adequate relief from postoperative pain.

Additionally, if pain is not promptly managed after surgery, it can hinder a patient's ability to walk, potentially causing adverse effects such as thromboembolism, myocardial ischemia, and arrhythmia.

The opioid analgesics are most commonly used as parenteral agents to manage post operative pain but the problem of respiratory depression remains to be considered.

This study is designed to compare the analgesic effect between dexmedetomidine versus magnesium sulfate as adjuvant to bupivacaine using ultrasound guided Transversus Abdominis Plane block in patients undergoing abdominal hysterectomy

DETAILED DESCRIPTION:
In addition to parenteral opioids and NSAIDS, various other methods used for post operative analgesia are infiltration of local anaesthetic agents, dermal patches, patient-controlled analgesia and epidural catheters, etc.

Numerous studies have demonstrated that when enhanced recovery procedures (ERPs) are used, hospital length of stay, time to return to normal function, postoperative ileus duration, thromboembolic complications, morbidity, and all of these factors are all reduced. In order to achieve the best pain treatment, many ERPs use a multimodal approach, decreasing the use of opioids as the primary analgesic in Favor of neuraxial and regional anaesthetic techniques.

One of the regional techniques routinely used is the transversus abdominis plane (TAP) block. Its widespread use in abdominal surgeries is due to its technical simplicity and trustworthy analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification I-ll,
* Aged >18 years,
* weight 50-85 kg,
* Patients who will undergo total abdominal hysterectomy

Exclusion Criteria:

* • ASA classification I-ll,

  * Aged >18 years,
  * weight 50-85 kg,
  * Patients who will undergo total abdominal hysterectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
the time of the first request of rescue analgesia | 24 hours
  the time of the first request of rescue analgesia (calculated from the time of the TAP block application)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu N, Long X, Lujan-Hernandez JR, Succar J, Xin X, Wang X. Transversus abdominis-plane block versus local anesthetic wound infiltration in lower abdominal surgery: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2014 Dec 15;14:121. doi: 10.1186/1471-2253-14-121. eCollection 2014. PMID 25580086